CLINICAL TRIAL: NCT02642861
Title: Cyclobenzaprine Treatment for Muscle Cramps in Cirrhotic Patients
Brief Title: Cyclobenzaprine in Muscle Cramps With Liver Cirrhosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Consultant liver and GIT diseases- Tanta university hospital, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Muscle cramps treatment
Record Dates: First submitted 2015-12-25; First posted 2015-12-30 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — cyclobenzaprine; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclobenzaprine (Active Comparator): Cyclobenzaprine administration for 2 weeks
  Interventions: Drug: Cyclobenzaprine
- PLacebo (Placebo Comparator): Calcium carbonate for 2 weeks
  Interventions: Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Cyclobenzaprine — cyclobenzaprine administration for 2 weeks
  Other Names: cyclosed
  Arms: Cyclobenzaprine
Drug: Calcium Carbonate — Calcium carbonate for 2 weeks
  Other Names: Calcitron
  Arms: PLacebo

SUMMARY:
- Cyclobenzaprine, is a muscle relaxer medication used to relieve skeletal muscle spasms. It is one of the best-studied drug for this application.

DETAILED DESCRIPTION:
Although a number of mechanisms for cramps in liver disease have been postulated and have been targeted by medical therapies, a clear picture of the causal events has not emerged. Several agents as vitamin E, human albumin, zinc, taurine, eperisone hydrochloride and branched-chain amino acids have shown some benefit in small uncontrolled studies, although large randomized controlled trials are lacking.

- Cyclobenzaprine, is a muscle relaxer medication used to relieve skeletal muscle spasms. It is one of the best-studied drug for this application.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis and has frequent muscle cramps

Exclusion Criteria:

* Allergy to cyclobenzaprine
* Encephalopathy.
* Receiving antidepressant drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of muscle cramps | 3 months
  The number of muscle cramps

CONTACTS AND LOCATIONS:
Overall Officials: Sherief M. Abd-Elsalam, Consultant, Principal Investigator — liver diseases dept.- Tanta university hospital; Walaa A. Elkhalawany, Consultant, Study Director — liver diseases dept.- Tanta university hospital
Locations (1):
- Tanta university - faculty of medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided